CLINICAL TRIAL: NCT03819777
Title: Volatile Organic Compounds as a Biomarker in Immune-mediated Pulmonary Arterial Hypertension
Brief Title: Volatile Organic Compounds (VOCs) as a Biomarker in Immune-mediated Pulmonary Arterial Hypertension (PAH)
Acronym: VOC-PAH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL57351.068.17
Record Dates: First submitted 2018-09-05; First posted 2019-01-29 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Pulmonary Arterial Hypertension; Systemic Sclerosis; Systemic Lupus
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood exhaled air
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Idiopathic PAH
- CTD-PAH
- CTD without PAH

SUMMARY:
Aim: to investigate the role of inflammation and auto-immunity in pulmonary arterial hypertension by using the profile of volatile organic compounds.

Hypothesis: first, the investigators hypothesize that at time of diagnosis the VOC profiles will discriminate patients with PAH-CTD and idiopathic PAH (IPAH) from patients with systemic sclerosis or systemic lupus erythematosus (CTD) without PAH, supporting the contention that there is a overlapping inflammatory and auto-immune pathway in PAH. During follow-up, the investigators will measure the VOC profiles of patients in all three groups who will be treated according standard clinical care. The hypothesis is that VOC profiles are affected by therapy.

ELIGIBILITY:
Inclusion Criteria:

1. PAH-CTD patients, inclusion criteria:

   * classification as definite systemic sclerosis or systemic lupus erythematosus according to respectively the ACR-EULAR criteria (16) and SLICC criteria (17)
   * minimal age of 18 year
   * diagnosis of pulmonary arterial hypertension: mean pulmonary artery pressure (mPAP) of ≥25 mmHg, pulmonary capillary wedge pressure (PCWP) ≤15 mmHg, and a pulmonary vascular resistance (PVR) ≥240 dynes.s.cm-5 measured by right heart catherization.
2. IPAH patients, inclusion criteria:

   * diagnosis of pulmonary arterial hypertension: mean pulmonary artery pressure (mPAP) of ≥25 mmHg, pulmonary capillary wedge pressure (PCWP) ≤15 mmHg, and a pulmonary vascular resistance (PVR) ≥240 dynes.s.cm-5 measured by right heart catherization.
   * no family history of PAH
   * triggering factor is excluded: connective tissue disease, drugs or toxins, human immunodeficiency virus, congenital heart disease, portal hypertension, schistosomiasis (2)
   * minimal age of 18 year
3. SSc and SLE (CTD) patients without PAH, inclusion criteria:

   * classification as definite systemic sclerosis or systemic lupus erythematosus according to respectively the ACR-EULAR criteria (16) and SLICC criteria (17)
   * minimal age of 18 year
   * no signs of PAH at screening visit

Exclusion Criteria:

* active or treated malignancy
* tuberculosis or hepatitis B/C infection in case of start immunosuppressive therapy
* need to start immediately with therapy
* already use of immune suppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Determining unique inflammatory VOC profiles in exhaled air in three groups of patients: IPAH, PAH-CTD and CTD without PAH. | 3 measurements in 2 weeks
  Exhaled air samples will be analyzed on inflammatory VOC profiles in the diagnostic phase of the study. Three measurements over a period of two weeks will be done. Statistically analysis will report one average VOC profile of the three measurements.
  Procedure: the patient is asked to exhale via a sterile mask into the ReCIVA breath sampler (Owlstone Medical, Cambridge, UK) in which mixed total exhaled air is immediately trapped and stored onto stainless-steel two-bed sorption tubes, filled with carbograph 1TD/Carbopack X (Markes International, Wales, UK). The tubes will be analyzed with GC-TOF-MS for the presence of VOCs after which multivariate statistical analysis will be used to select those VOCs unique for the various patient groups.

SECONDARY OUTCOMES:
Correlation between unique inflammatory VOCs to well-established biomarkers of immune activation and inflammation in PAH-CTD and idiopathic PAH. | 1 measurement at baseline
  The correlation analysis by means of bivariate (Spearman correlation) and multivariate analysis (canonical correlation analysis) will be performed.
Change (Δ, delta) from baseline in selective inflammatory VOC profiles after 3, 6 and 12 months in all patients treated with PAH and/or immunsuppressive medication. | Changes (Δ, delta) between baseline, 3 months, 6 months, 9 months and 12 months
  Wilcoxon signed-rank test will be utilized to see if the individual, selective inflammatory VOCs after treatment significantly differ with the baseline measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Pieter van Paassen, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided